CLINICAL TRIAL: NCT03040115
Title: Assessment of Safety of Air Travel in Patients With Birt-Hogg-Dube Syndrome
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nishant Gupta, MD, MS, Adjunct Assistant Professor, University of Cincinnati
Other Study IDs: RLDC5714A; U54HL127672 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-02-02 (Estimated); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Birt-Hogg-Dube Syndrome
MeSH Terms: conditions — Birt-Hogg-Dube Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Non-Interventional Study

SUMMARY:
The aim of this study is to conduct survey-based assessments for the safety of air travel in patients with Birt-Hogg-Dube syndrome (BHD). The study will enroll patients through the clinic network at Rare Lung Disease Consortium (RLDC) and through the BHD foundation website. Patients will have access to the questionnaire via REDCap (an online data management system) and each patient will be provided with a link to complete the survey. The investigators plan on enrolling approximately 100 patients with BHD for the purpose of this study. Secondary aims of this study include further characterization of the clinical aspects of disease and to establish a contact registry for these patients, in order to facilitate future studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 or older
* English literate
* Signed, dated informed consent; either given electronically or via paper form
* Diagnosis of BHD confirmed by either a) the presence of fibrofolliculomas/trichodiscomas on skin biopsy, or b) the presence of pathogenic FLCN mutations.

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of Birt-Hogg-Dube syndrome are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Gupta, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Self-reporting With BHD: Patients self-reporting with BHD
Period: Overall Study
Arm/Group | Patients Self-reporting With BHD
Started | 104
Completed | 104
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Self-reporting With BHD
Number analyzed (Participants) | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at time of survey collection
  years | 50 [39 to 61]
Sex: Female, Male [Count of Participants; unit: Participants] — Patients self-reported gender.
  Participants
    Female | 86
    Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104
Number of Participants with a History of Air Travel [Number; unit: participants] | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Birt-Hogg-Dube Syndrome Who Experienced Spontaneous Pneumothorax During or Within 24 Hours Following Air Travel
Description: The investigators will measure the number of pneumothoraces that occur either during air travel, or within 24 hours of air travel among patients with Birt-Hogg-Dube syndrome. The incidence of air travel related pneumothorax will be calculated by dividing the number of pneumothoraces to the total number of flights undertaken by the entire cohort.
Time Frame: During air travel or within 24 hours following air travel
Measure: Count of Participants; unit: Participants
Groups:
- BHD Patients With Air Travel Related Pneumothorax: Air travel related pneumothorax in patients with BHD
Arm/Group | BHD Patients With Air Travel Related Pneumothorax
Number analyzed (Participants) | 104
Participants | 8

2. Secondary Outcome: Number of Patients With Birt-Hogg-Dube Syndrome Who Experience a Spontaneous Pneumothorax
Description: The investigators will catalogue the number of spontaneous pneumothoraces experienced by patients with Birt-Hogg-Dube syndrome.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- Patients With BHD Related Spontaneous Pneumothorax: Patients self-reporting spontaneous pneumothorax associated with BHD
Arm/Group | Patients With BHD Related Spontaneous Pneumothorax
Number analyzed (Participants) | 104
Participants | 79

3. Secondary Outcome: Number of Patients With Birt-Hogg-Dube Syndrome Who Experience Recurrent Pneumothorax Following Pleurodesis
Description: The investigators will measure the incidence of ipsilateral pneumothorax following pleurodesis in order to determine the efficacy (as measured by the rate of pneumothorax recurrence following pleurodesis).
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- BHD Patients With Recurrent Pneumothorax Following Pleurodesis: Number of patients with Birt-Hogg-Dube syndrome who experience recurrent pneumothorax following pleurodesis
Arm/Group | BHD Patients With Recurrent Pneumothorax Following Pleurodesis
Number analyzed (Participants) | 79
Participants | 29

ADVERSE EVENTS:
Time Frame: Not applicable. Cross sectional study.
Description: Cross sectional study. No data regarding mortality, serious or other adverse events was collected as part of the study.
Groups:
- EG000: AEs were not collected as part of this observational study.
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03040115/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT03040115/SAP_001.pdf
  • Informed Consent Form (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03040115/ICF_002.pdf